CLINICAL TRIAL: NCT00356616
Title: Open-Label, Single-Centre, Randomised Pilot Study to Evaluate Immunovirological and Clinical Evolution of a Combination With Nucleoside Analogues/Nucleotides (Trizivir +Tenofovir) in Multiresistant Patients With Virological Failure
Brief Title: Immuno-Virological Efficacy of Combination With Trizivir +Tenofovir in Multiresistant HIV Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Lluita Sida Foundation, Lluita Sida Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TETRIZ; 2005-002203-17
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2007-11

CONDITIONS: HIV Infections
Keywords: Antiretroviral treatment; virological failure; HIV
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine, and zidovudine drug combination; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Trizivir+ Tenofovir 2/day
  Interventions: Drug: Trizivir (AZT+3HT+Abacavir) twice daily; Drug: Viread (300 mg Tenofovir disoproxil fumarate) once daily
- B (No Intervention): antiretroviral treatment optimizated by genotyp

INTERVENTIONS:
Drug: Trizivir (AZT+3HT+Abacavir) twice daily — Trizivir (AZT+3HT+Abacavir) twice daily
  Arms: A
Drug: Viread (300 mg Tenofovir disoproxil fumarate) once daily — Viread (300 mg Tenofovir disoproxil fumarate) once daily
  Arms: A

SUMMARY:
To evaluate whether the combined therapy of two nucleosides plus one nucleotide (Trizivir + TDF) manages to keep CD4 lymphocytes stable in patients with HIV infection on antiretroviral treatment that present virological failure and multiple resistance to antiretrovirals.

DETAILED DESCRIPTION:
This study has been designed to determine whether the use of a regimen based exclusively on NTRI, containing tenofovir, zidovudine and lamivudine, is able to preserve immunological status in patients with detectable viral load for whom an efficacious salvage regimen cannot be designed, slowing the progression of the viral load and reducing antiretroviral treatment-associated toxicity. In order to complete the salvage regimen without increasing the number of tablets too much, Trizivir plus tenofovir as investigational treatment will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Age>= 18 years.
2. HIV-1 infected patients.
3. Patients on antiretroviral treatment including NTRI + PI +/- NNRTI +/- fusion inhibitors at inclusion in the study.
4. Virological failure, defined as 2 determinations with viral load >1,000 copies/mL in the last 6 months, during stable HAART therapy over the previous 6 months.
5. Genotype or phenotype resistance to three families of antiretrovirals (PI, NTRI and NNRTI) demonstrated in genotype study carried out in the last 48 weeks and defined as:

   * 3 or more TAMS of the following: M41L, E44D, D67N, V118I, L210W, T215Y/F, K219Q/E.
   * Existence of the M184V mutation or probable presence in the cellular archives.
   * 5 or more mutations that confer resistance to PI of the following: I10F/I/R/V, V32I, M46I/L, I54V/M/L, V82A/F/T/S/V, I84V/A/C, L90M.
   * Existence of 1 or more mutations that confer resistance to NNRTI, or probable presence in the cellular archives of: K103N, Y181C/I/Y, G190S/A/G.
6. CD4 lymphocytes >- 300 cells/mm3 in the last two determinations.
7. Subject able to follow the treatment period.
8. Acceptance of the study and signature of the informed consent form.
9. Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use a barrier contraceptive method during the study.

Exclusion Criteria:

* Suspicion of previous incorrect adherence.
* Pregnancy or breastfeeding
* Suspicion of intolerance to any investigational drug.
* Record of any disease which, according to clinical criteria, may reoccur with the proposed change of therapy (sarcoma, lymphoma, etc).
* CD4 Nadir below 200 cel/mm3.
* Acute intercurrent disease or fever in the 15 days before inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Variations in the immune status of patients in each group throughout follow-up. | 48 weeks

SECONDARY OUTCOMES:
Percentage of patients that increase viral load by > 0.5 log | weeks 12, 24, 36 and 48
Percentage of patients that increase viral load by > 100,000 copies/mL | weeks 12, 24, 36 and 48
Percentage of patients that present some clinical event, B or C classification according to the CDC. | during the 48 weeks of follow-up
Percentage of patients that present clinical or analytical adverse effects degree > 2 according to the WHO classification. | weeks 12, 24, 36 and 48
Percentage of patients that drop out of treatment. | weeks 12, 24, 36 and 48
Percentage of patients that drop out of the study due to intolerance or adverse effects. | weeks 12, 24, 36 and 48
Percentage of change in lipid determinations. | weeks 12, 24, 36 and 48 with regard to baseline
Percentage of patients that report changes, improvement or worsening in redistribution of body fat. | weeks 12, 24, 36 and 48
Percentage of patients that present adherence to the antiretroviral treatment > 95%. | weeks 12, 24, 36 and 48
Percentage of patients that present improvement in the quality of life (MOS-HIV) and satisfaction questionnaires. | weeks 12, 24, 36 and 48
Percentage of patients that present an increase in the number of active drugs. | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unit
Locations (1):
- H.U. Germans Trias i Pujol, Badalona, Barcelona, Spain